CLINICAL TRIAL: NCT01963559
Title: Cutaneous Microcirculation and Diabetic Foot
Acronym: M2P2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011.661
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Diabetic Foot Proned Patients
MeSH Terms: interventions — Lidocaine; Prilocaine; Administration, Topical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetic patients with MPP (Other)
  Interventions: Drug: Lidocaine/prilocaine 1g (topical administration)
- Diabetic patients without MPP (Other)
  Interventions: Drug: Lidocaine/prilocaine 1g (topical administration)

INTERVENTIONS:
Drug: Lidocaine/prilocaine 1g (topical administration) — Cutaneous blood flow measurement using laser Doppler

SUMMARY:
15% of diabetics have a diabetic foot (DF) in their lives associated with a risk of amputation and mortality two times greater than that of a diabetic population without DF. Predicting the occurrence of an DF is limited and only the occurrence of a diabetic wound up involved assessment and treatment. Our team is behind the discovery of the Pressure-Induced Vasodilation (PIV) first observed in healthy subjects after local application of a gradual pressure on the skin leading to cutaneous vasodilation at the application of pressure. This gain in blood flow delays the onset of ischemia. However the involvement of PIV in the DF, which is also a pressure-induced skin lesion, remains to be demonstrated in diabetic subjects. The main objective of this study is to show that PIV, a functional examination of the cutaneous microcirculation we developed, is altered in the presence of DF, taking into account the influence of age and neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Adult Men and Women
* Presence of diabetes
* Signed acknowledgement form

Exclusion Criteria:

* No signed acknowledgement form
* patients under 18 year-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Cutaneous blood flow | Within 3 months after inclusion

SECONDARY OUTCOMES:
Effect of neuropathy on PIV impairment | Within 3 months after inclusion
  Difference in skin vascular response to local application of pressure (PIV) with and without topical application of a local anesthetic cream Lidocaine / prilocaine in all diabetic patients (with and without MPP).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite, France